CLINICAL TRIAL: NCT06852703
Title: Predictive BioMArkers of AlTERed NeurologicAL Trajectories Consequent to PrenataL
Brief Title: Predictive BioMArkers of AlTERed NeurologicAL Trajectories Consequent to PrenataL InflammatorY Insults
Acronym: MATERNALLY
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Sponsor
Other Study IDs: ID 18657
Record Dates: First submitted 2024-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Biomarkers; Neurodevelopmental Disorders; Inflammation, Brain
MeSH Terms: conditions — Neurodevelopmental Disorders; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: healthy mothers
- diseased: Infected mothers
  Interventions: Other: Infection during pregnancy

INTERVENTIONS:
Other: Infection during pregnancy — any bacterial or viral infection acquired during pregnancy
  Groups: diseased

SUMMARY:
Inflammation during pregnancy represents an important risk factor for the development of neuropsychiatric disorders in the offspring. Despite clear epidemiological data supporting this association, translational studies aimed at identifying early predictive biomarkers and possible interventional strategies for this pathological condition are still missing. The MATERNALLY proposal aims to assess in a large patient cohort a novel multiparametric approach for the identification of predictive postnatal behavioral and circulating biomarkers. In parallel, a controlled mouse model for maternal immune activation will be exploited to understand the basic molecular mechanism that links inflammation with aberrant neural circuit formation and to unveil possible therapeutic targets. The integration of the two approaches will allow identifying early predictive biomarkers and proof of principle interventional strategies for this condition of high practical relevance to the neonatologist community

DETAILED DESCRIPTION:
This is a pilot study that will assess 300 mothers and an equal number of children. Patients will be recruited until the predetermined sample size is reached at the Department of Obstetrics and Gynecology I, University Hospital of Pisa, by the team coordinated by Prof. Simoncini.

All children will be followed for the first year of life by the team at the IRCCS Fondazione Stella Maris in Pisa, coordinated by Prof. Guzzetta.

Study on mothers The presented study involves the use of biological samples and fetal ultrasound evaluations performed at various stages of pregnancy.

The recruitment will involve 300 pregnant women at 11-14 weeks of gestation: recruitment will take place in the first trimester during access to the Department of Obstetrics and Gynecology I University Hospital for the execution of first-trimester screening ultrasound (combined test) as per clinical practice.

The biological samples will consist of whole blood samples useful for dosing the circulating levels of IL-6, PCR, PCT, TSH, and vitamin D, which are beyond the routinely screened parameters in pregnancy: collection will be performed in the first, second, and third trimesters with the aim of obtaining a longitudinal immunological profile throughout the pregnancy.

Maternal biological samples will be collected as four additional aliquots (IL 6- 6 cc, PCR and PCT - 6 cc, TSH - 6 cc, 25-OH Vit D -6 cc for a total of 24 cc) during the routine sampling planned by the approved pathway by the SSN:

The first sampling will take place during the combined test, i.e., at the time of enrollment at the Department of Obstetrics and Gynecology I, where a blood sample is planned for the measurement of PAPP-A and free-beta-HCG (as per screening for chromosomal abnormalities); The second sampling will be performed concurrently with the first ultrasound assessment planned by the study and, in Toxo-test negative patients, may coincide with the performance expected from the pregnancy booklet; The third sampling will be performed concurrently with the third ultrasound assessment planned by the study and may coincide with the performance expected from the pregnancy booklet (third-trimester infectious screening);

Samples taken at the Department of Obstetrics and Gynecology I will be processed and analyzed as follows:

Samples for TSH and 25-OH Vit D will be sent to the Laboratory of Chemistry and Endocrinology (Cisanello Establishment Ed. 8 Director Dr. Maria Rita Sessa) Samples for IPCR and PCT will be sent to the Laboratory of Clinical Chemical Analysis (Santa Chiara Establishment Director Dr. Giovanni Pellegrini) The sample for IL-6 will be sent to the Laboratory of Clinical Pathology (Santa Chiara Establishment Director Dr. Paolicchi) The costs of such extra-routine determinations will be fully covered by the funds made available for the study in question.

Samples will be sent on the same day of collection to the laboratories with specific competence which will handle the processing of the blood sample and subsequent disposal according to their specific operating protocol.

Ultrasound examinations will be obtained by obtaining additional scans during the obstetric ultrasound screenings in the second (between 20 and 21 weeks of gestation) and third trimesters (30-31 weeks of gestation) respectively.

The ultrasound assessment includes:

Sonographic study of the CNS, which involves the following anatomical-biometric evaluations:

Visualization of the midline and the cavity of the septum pellucidum Visualization of the corpus callosum and measurement of the anteroposterior diameter in sagittal section Visualization of the 3rd and 4th cerebral ventricles Visualization and measurement of both lateral ventricles (latero-lateral diameter) Morphological and dimensional evaluation of the cerebellar vermis Visualization of the cerebellar hemispheres Measurement of the transcerebellar diameter (TCD) Measurement of the anteroposterior diameter of the cisterna magna Morphological and dimensional evaluation of the cerebral hemispheres, the Sylvian fissure, the insular lobe, and the parieto-occipital fissure Dimensional evaluations will be compared to specific reference tables for gestational age.

Morphological evaluations will establish regular/irregular morphology for the gestational age reference

Evaluation of the number of major fetal movements according to specific score, throughout the duration of the ultrasound examinations (approximately 30 minutes), in particular:

Movements of the upper and lower limbs (flexion-extension) Sucking Swallowing Change of position (longitudinal or transverse) or presentation (cephalic, podalic) Respiratory movements Ultrasound assessments will be performed in the prenatal diagnosis clinics of the AOUP Obstetrics and Gynecology in Pisa Ed. 2 and Ed.5 Santa Chiara. The equipment used is the Samsung WS80A ultrasound system product code USS-WS8AL44/WR, provided at the main investigator's affiliated institution.

Follow-up procedure for children born to mothers enrolled in the study:

Evaluation of spontaneous movements (General Movements - GMs): This is an assessment of the quality of spontaneous movements and is one of the most sensitive and specific tests for the diagnosis of Infantile Cerebral Palsy. An initial assessment will take place in the first days of life at the neonatology unit of Santa Chiara Hospital in Pisa, before discharge. Subsequent evaluations will be obtained via video recording every two weeks, by the child's parents, in a home environment. Video recordings will stop when the child reaches 20 weeks of corrected age, as during this period spontaneous motor activity disappears and voluntary motor activity emerges. Parents will be extensively explained how to perform the assessment and what it consists of.

Magnetic Resonance Imaging (MRI) - on 50 newborns. The MRIs will be performed at the IRCCS Fondazione Stella Maris on newborns of 6 weeks corrected age whose mothers, at the time of obtaining informed consent, have agreed to undergo the examination. Once the number of 50 newborns who have undergone Magnetic Resonance Imaging (MRI) is reached, it will not be necessary to continue with the execution of the examination, as it is no longer useful for the purposes of the study.

The MRIs will be performed on newborns of 6 weeks corrected age, during spontaneous sleep. Cortical thickness, volumes and gyrification, connectivity, and CBF measures will be modeled as a function of inflammatory indicators through both linear and nonlinear models. Voxel-wise linear and nonlinear regression models will be used to assess changes in MRI considering postmenstrual age, sex, maternal inflammatory levels, and neonatal motor activity.

Motor outcome: The motor outcome of the children of the mothers participating in the study will be assessed at one year of corrected age, using the standardized scale The Alberta Infant Motor Scale (AIMS). This is an assessment scale of gross motor development in children from birth until they achieve independent walking. The AIMS includes 58 items organized into four positions: prone, supine, sitting, and standing. Each item describes three aspects of motor performance: load movements, postures, and antigravity movements. Abnormal results obtained on the Alberta Infant Motor Scale predict pathological motor outcome in 86% of cases

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 40 years. BMI between 18 kg/m2 and 25 kg/m2. Negative remote medical history for chronic conditions (rheumatological, immunological, endocrinological).

Negative obstetric history for significant pathologies (pre-eclampsia, gestational diabetes, preterm birth).

Reassuring combined test

Exclusion Criteria:

* Pre-gestational diabetes
* Multiple pregnancy
* Threatened preterm labor and/or premature rupture of membranes
* Pre-eclampsia
* Intrauterine growth restriction (IUGR)
* Fetal macrosomia (biometrics >90th percentile)
* Chromosomal syndromes, genetic conditions, or multiple fetal malformations or major fetal malformations
* Withdrawal of informed consent
* Smoking patients are not excluded from the study, nor are patients who develop gestational diabetes during pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Not applied
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers analysis on blood samples collected from healthy and infected mothers | 32 month
  Assesment of the immune profile in both cohorts recruited. In particular, we will measure the circulating levels of IL-6, CRP, PCT, TSH and Vitamine D at 20 and 30 weeks gestation to obtain a longitudinal immune profile across gestation. The analysis will be carried out using ELISA kit in the serum collected from both cohorts.
Sonographic examination at fetal level | Once during the second and the third trimester of pregnancy
  Brain ultra-sound study involves axial, coronal and sagittal planes to obtain qualitative anatomic parameters related to Head shape, Integrity of falx cerebri,, Cavum septum pellucidum, Thalami, Insulae lobes, Cerebral hemispheres, Third and fourth ventricles, Parieto-occipital fissure
Sonographic examination at fetal level | Once during the second and the third trimester of pregnancy
  Brain ultra-sound study involves axial, coronal and sagittal planes to obtain quantitative anatomic parameters related to (in mm) Head circumference and biparietal diameter (axial plan), Antero-posterior diameter of corpus callosum (sagittal plan), Cerebellum (axial plan), Cerebellar vermis, cranio-caudal diameter (sagittal plan), Lateral ventricles, latero-lateral diameter (axial plan), Cisterna magna, antero-posterior diameter (axial plan)
Sonographic examination at fetal level | Once during the second and the third trimester of pregnancy
  Brain ultra-sound study involves axial, coronal and sagittal planes to obtain quantitative anatomic parameters (in angle) related to Sylvian fissure (coronal plan)
Sonographic examination at fetal level | Once during the second and the third trimester of pregnancy
  Quantitative and qualitative evaluation of fetal movements including, Flexion and extension of fetal of arms or legs, Sucking movements, Swallowing movements, Situation changes (longitudinal or trasversal) or presentation changes (cephalic, breech), Breathing movements
Newborns: assessment of spontaneous movements | 3 times between birth and 20 weeks post-term
  Assessment of spontaneous movements based on Prechtl method of general movements assessment. From longitudinal videorecordings performed by the parents in a structured home setting, we will assess the GM optimality score. The scale between 0 and 38 points from 0-9 weeks post-term; and 5-28 points from 10-20 weeks post-term. A lower score means poorer predicted motor outcome
Infant behavioral and motor assessment | 12 months infant age
  Infant behavioral and motor assessment according to Alberta Infant Motor Scale. The scale is between 0 and 58 points. A lower score on the Alberta Infant Motor Scale (AIMS) indicates delayed or less advanced motor development

SECONDARY OUTCOMES:
Newborns: Magnetic resonance imaging (MRI) | Once between birth and 8 weeks infant age
  Magnetic resonance imaging (MRI) will be performed while the participant is in natural sleep to assess brain structure and function. The following parameters will be measured:
  Cortical Thickness: Measured in millimeters (mm); higher values indicate thicker cortex.
Newborns: Magnetic resonance imaging (MRI) | Once between birth and 8 weeks infant age
  Magnetic resonance imaging (MRI) will be performed while the participant is in natural sleep to assess brain structure and function. The following parameters will be measured:
  Volumes: Measured in cubic millimeters (mm³) for brain regions; larger volumes may indicate more developed structures
Newborns: Magnetic resonance imaging (MRI) | Once between birth and 8 weeks infant age
  Magnetic resonance imaging (MRI) will be performed while the participant is in natural sleep to assess brain structure and function. The following parameters will be measured:
  Gyrification: Quantified as a gyrification index (dimensionless ratio); higher values reflect more cortical folding.
Newborns: Magnetic resonance imaging (MRI) | Once between birth and 8 weeks infant age
  Magnetic resonance imaging (MRI) will be performed while the participant is in natural sleep to assess brain structure and function. The following parameters will be measured:
  Connectivity: Measured using structural metrics: fractional anisotropy and mean diffusivity.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUP, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No